CLINICAL TRIAL: NCT07193134
Title: Genetically Modified Epidermolysis Bullosa Self-Assembled Skin Substitute (GMEB-SASS) to Treat Patients Suffering From Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: GMEB-SASS: A Gene-Modified Skin Substitute for RDEB Treatment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOEX 020; 291541 (Other: Health Canada)
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: RDEB; Recessive Dystrophic Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica, Recessive
Keywords: Skin Abnormalities; Congenital Abnormalities; Epidermolysis Bullosa; Skin Diseases, Genetic; Genetic Diseases, Inborn; Collagen Diseases; Connective Tissue Diseases; Skin and Connective Tissue Diseases; Skin Diseases; Skin Diseases, Vesiculobullous; Epidermolysis Bullosa Dystrophica; Genetic therapy; Autologous Skin Graft; SIN Retroviral Vector; Type VII Collagen; COL7A1
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Skin Abnormalities; Congenital Abnormalities; Epidermolysis Bullosa; Skin Diseases, Genetic; Genetic Diseases, Inborn; Collagen Diseases; Connective Tissue Diseases; Skin and Connective Tissue Diseases; Skin Diseases; Skin Diseases, Vesiculobullous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMEB-SASS (Experimental): All patients will receive GMEB-SASS
  Interventions: Drug: Genetically Modified Epidermolysis Bullosa Self-Assembled Skin Substitute (GMEB-SASS)

INTERVENTIONS:
Drug: Genetically Modified Epidermolysis Bullosa Self-Assembled Skin Substitute (GMEB-SASS) — Wound debridement will be performed, followed by the application of temporary allogeneic skin grafts for 3-5 days. The allografts will then be removed, and the GMEB-SASS grafts will be applied.

SUMMARY:
This study is being done to find out if a new type of skin graft, called GMEB-SASS, is safe and effective for helping wounds heal in people with RDEB (Recessive Dystrophic Epidermolysis Bullosa).

The GMEB-SASS graft contains two types of living skin cells: keratinocytes and fibroblasts. It is made in a laboratory using a small sample of the patient's own skin.

To help the patient's skin cells produce a missing protein called type VII collagen, scientists grow the patient's cells in the lab and use a virus-like tool (called a retroviral vector) to give the cells the correct instructions. This allows the cells to make the normal protein that is missing in people with RDEB.

The graft is designed to be permanent, and the goal is to improve wound healing by replacing damaged skin cells with healthy ones.

DETAILED DESCRIPTION:
The GMEB-SASS is a skin tissue composed of living cells genetically modified in the laboratory to express a functional form of type VII collagen. The GMEB-SASS integrates with the patient's skin once grafted. The graft is autologous and expected to be permanent.

This is a first-in-human trial aiming to explore indications of the safety and efficacy of the GMEB-SASS skin graft in healing skin wounds in RDEB patients. Adults and children are included. However, a risk mitigation measure was added in order that at least some safety data from adults be available before the pediatric population is treated. Therefore, the study design is adaptative and divided into two phases: a learning phase (phase A) and a confirmatory phase (phase B).

In the present trial, the investigators hypothesize that retroviral transfer of the COL7A1 gene, combined with the use of the self-inactivated (SIN) COL7A1 vector, will restore a functional dermo-epidermal junction in the bilayer tissue-engineered skin produced at the LOEX research center by the self-assembly method. The method for the production of substitutes is similar to the one used in the ongoing clinical trial for the treatment of burn patients (ClinicalTrials.gov Identifier: NCT02350205) using SASS, with the exception of gene modification.

An important issue in RDEB patients is that their skin is colonized by bacteria due to the continuous presence of wounds. The method used to decontaminate the graft bed is crucial to ensure proper integration of the GMEB-SASS. The proposed intervention in this trial involves two surgical steps: the use of allografts to prepare the graft bed in a first step, followed by the application of the GMEB-SASS a few days later. This approach will be applied to at least participants enrolled in Phase A of the study.

The maximum daily dose per grafting session is the number of GMEB-SASS covering a maximum of 9% of the total body surface area. The number will be calculated based on the participant's height, weight, and age.

ELIGIBILITY:
Inclusion Criteria:

* Age

Learning phase:

* Subjects 1 to 3: Eighteen (18) years old or older.
* Subjects 4 to 6: Twelve (12) years old or older.
* Subjects 7 to 9: Seven (7) years old or older.

Other Inclusion Criteria:

* Clinical diagnosis of recessive dystrophic epidermolysis bullosa (RDEB) with confirmed biallelic pathogenic variant in the COL7A1 gene.
* Candidates - or their parents/caregivers if the candidates have limited comprehension, who are able to understand the study and to comply with the study procedures.
* On the day of grafting, one or more blistered and/or erosive skin areas on the trunk and/or extremities large enough to graft at least three 25 to 50 cm2 GMEB-SASS grafts.
* Ability to undergo anesthesia.

Exclusion Criteria:

* Medical instability limiting the ability to travel to the investigative center.
* Any medical condition or illness that may impact study participation or compromise the safety of the participants, as per the investigator's judgment.
* Evidence of systemic infection.
* Current evidence or a history of non-metastatic or metastatic squamous cell carcinoma at the site to be grafted.
* Any clinically significant abnormal laboratory values or abnormal findings identified during physical examination or through medical history that could compromise participant safety, as per the investigator's judgment.
* History of or known allergy to bovine proteins.
* Active drug or alcohol addiction.
* Female candidate who are pregnant or breast-feeding.
* Candidate who has received immunotherapy, including oral corticosteroids (Prednisolone > 1 mg/kg), for more than one week, within 2 weeks prior to the study intervention (initial biopsy and GMEB-SASS grafting) (intranasal and topical preparations are permitted).
* Candidate who has received chemotherapy within 60 days prior to the study intervention (initial biopsy and GMEB-SASS grafting).
* Candidate who has received, in the last 6 months prior to the study intervention (initial biopsy and GMEB-SASS grafting), any gene therapy, chemical or biological product modifying collagen 7 expression.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 12 months
  Record of Adverse Events (AE), Serious Adverse Events (SAEs), Adverse Reactions (ARs) and Serious Adverse Reactions (SARs).
Pain score changes using a Visual Analogue Scale (VAS) | Baseline, week 2, months 1, 3, 6 and 12
  Pain score of the grafted wounds for the past 7 days. Horizontal line, typically 10 centimeters in length, anchored by two verbal descriptors: 0 = No pain; 10 = Worst pain possible.
Itch score changes using a Visual Analogue Scale (VAS) | Baseline, week 2, months 1, 3, 6 and 12 post intervention
  Itch score of the grafted wounds for the past 7 days (100-point visual analog scale). Horizontal line, typically 10 centimeters in length, anchored by two verbal descriptors: 0 = No itch, 100 = Worst itch Time Frame: Baseline, week 2, months 1, 3, 6 and 12

SECONDARY OUTCOMES:
Percentage of the grafted GMEB-SASS surface area that has healed | Week 2, months 1, 3, 6 and 12 post intervention
  Percentage of epithelialization
iscorEB questionnaire - clinician portion | Baseline, months 3 and 12 post intervention
  Instrument for scoring clinical severity outcomes for research of EB. iscorEB is a measurement tool for evaluating the disease severity in EB patient. It evaluates the cutaneous, mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. Score ranges between 0-138 for the clinician subscore.
Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) | Time Frame: Baseline, months 3 and 12 post intervention
  Instrument for scoring clinical severity outcomes for research of EB. Total EBDASI activity score ranges of 0-42 (mild), 43-106 (moderate) and 107-506 (severe).

OTHER OUTCOMES:
Quality of Life Epidermolysis Bullosa (QOLEB) questionnaire | Baseline, months 1, 3, 6 and 12
  Instrument for scoring quality-of-life. 17 questions covering physical, emotional, and social aspects of living with EB, with four response choices from "not at all" to "constant".
Quality-of-life EQ-5D questionnaire | Baseline, months 1, 3, 6 and 12
  Tool developed by the EuroQol Group to measure health-related quality of life. It evaluates health across five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: from no problems to extreme/unable. The tool includes a visual analogue ccale (EQ VAS):
  a vertical scale from 0 ("worst health imaginable") to 100 ("best health imaginable") where patients rate their overall health.
Quality-of-life iscorEB questionnaire - patient portion | Baseline, months 1, 3, 6 and 12
  Instrument for scoring clinical severity outcomes for research of EB. It evaluates the cutaneous, mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. The patient portion of the iscorEB instrument, is considered a quality-of-life measure because it captures the patient's internal perceptions and experiences. Score ranges between 0-120 for the patient subscore.
Scar evaluation - Vancouver scar scale (VSS) | months 3, 6 and 12
  The Vancouver Scar Scale (VSS) is a tool used to measure scar severity across four aspects: vascularity (0-3), pliability (0-5), pigmentation (0-3), and scar height (0-4). The total score ranges from 0 (best outcome) to 15 (worst outcome).
Participant's self-perception about the persistence of healing in the treated areas | Months 3, 6 and 12
  The participant is asked about the durability of the GMEB-SASS under study compared with the skin before, choosing from three options: more durable (better), no change, or less durable (worse).
Participant's self-perception of how easily the skin blisters in the treated areas | Months 3, 6 and 12
  The participant is asked how easily the GMEB-SASS under study blister compared with the skin before, choosing from three options: more resistant to blistering (better), no change, blisters more easily (worse)
Type VII collagen protein expression | Baseline, months 3 and 12
  Type VII collagen protein expression in tissue biopsies
Autoantibody against type VII collagen | Baseline, month 3 post intervention if signs of rejection, month 12 for others
  Change in the level of autoantibody against type VII collagen in the blood
Economic impact evaluation | Baseline, months 1, 6, 12
  Economic impact evaluation questionnaire: tool to measure direct and indirect costs of a health condition for patients and their families.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Germain, PhD, Study Director — CHU de Québec-Université Laval; Elena Pope, MD, FRCPC, Principal Investigator — The Hospital for Sick Children (SickKids)
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No